CLINICAL TRIAL: NCT02109445
Title: PHASE 1/2 STUDY OF PF-03084014 IN COMBINATION WITH GEMCITABINE AND NAB-PACLITAXEL IN PATIENTS WITH PREVIOUSLY UNTREATED METASTATIC PANCREATIC DUCTAL ADENOCARCINOMA
Brief Title: Study Of PF-03084014 In Combination With Gemcitabine And Nab-Paclitaxel In Patients With Metastatic Pancreatic Adenocarcinoma Not Previously Treated With Anticancer Therapies
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated on 24JUN15 due to change in strategy of PF-03084014 development.No safety/efficacy concerns were behind the reason of trial termination
Sponsor: Pfizer (Industry)
Collaborators: Academic GI Cancer Consortium (AGICC) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: A8641019; 2013-005574-21 (EudraCT Number)
Record Dates: First submitted 2014-04-02; First posted 2014-04-09 (Estimated); Results first posted 2017-06-12 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2018-12

CONDITIONS: Metastatic Cancer Pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — nirogacestat; Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Phase 1 (Experimental): PF-03084014 in combination with gemcitabine and nab-paclitaxel
  Interventions: Drug: PF-03084014; Drug: Gemcitabine; Drug: Nab-paclitaxel
- Phase 2 Arm A (Experimental): PF-03084014 in combination with gemcitabine and nab-paclitaxel
  Interventions: Drug: PF-03084014; Drug: Gemcitabine; Drug: Nab-paclitaxel
- Phase 2 Arm B (Active Comparator): Gemcitabine plus nab-Paclitaxel
  Interventions: Drug: Gemcitabine; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: PF-03084014 — Tablets, orally administered twice daily on a continuous dosing schedule in 28 days cycles. Doses: 100 -150 mg BID
  Arms: Phase 1
Drug: Gemcitabine — Intravenously administered on Days 1, 8, 15 in 28 days cycles at the dose of 1000 mg/m2.
  Arms: Phase 1
Drug: Nab-paclitaxel — Intravenously administered on Days 1, 8, 15 in 28 days cycles at the dose of 125 mg/m2.
  Other Names: Abraxane
  Arms: Phase 1
Drug: PF-03084014 — Tablets, orally administered twice daily on a continuous dosing schedule in 28 days cycles. Phase 2 dose will be the recommended phase 2 dose defined in phase 1.
  Arms: Phase 2 Arm A
Drug: Gemcitabine — Intravenously administered on Days 1, 8, 15 in 28 days cycles at the dose of 1000 mg/m2.
  Arms: Phase 2 Arm A
Drug: Nab-paclitaxel — Intravenously administered on Days 1, 8, 15 in 28 days cycles at the dose of 125 mg/m2.
  Other Names: Abraxane
  Arms: Phase 2 Arm A
Drug: Gemcitabine — Intravenously administered on Days 1, 8, 15 in 28 days cycles at the dose of 1000 mg/m2.
  Arms: Phase 2 Arm B
Drug: Nab-paclitaxel — Intravenously administered on Days 1, 8, 15 in 28 days cycles at the dose of 125 mg/m2.
  Other Names: Abraxane
  Arms: Phase 2 Arm B

SUMMARY:
This study consists of a Phase 1b portion aimed to determine the maximum tolerated dose and the safety profile of PF-03084014 in combination with gemcitabine and nab-paclitaxel followed by a Phase 2 portion to evaluate the efficacy of the triple combination in terms of overall survival in patients with metastatic pancreatic ductal adenocarcinoma not previously treated with anticancer therapies.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically diagnosis of metastatic ductal adenocarcinoma of the pancreas.
* No prior radiotherapy, surgery chemotherapy or investigational therapy for metastatic disease. Prior adjuvant therapy with 5-FU or gemcitabine (± gemcitabine post radiation) administered as radiosensitizer allowed, provided at least 6 months have elapsed between the last dose and study registration
* Tumor tissue available (Archival 6 months old or de novo biopsy)
* Measurable disease as per RECIST 1.1
* Performance Status (ECOG) 0 or 1

Exclusion Criteria:

* Symptomatic brain metastases requiring steroids
* Prior therapy with gamma secretase inhibitors or other Notch pathway inhibitor
* Major surgery within 4 weeks of registration in the current study
* Known hypersensitivity to gemcitabine or nab-paclitaxel or any of the excipients
* Current or anticipated need for food or drugs that are strong/moderate CYP3A4 inhibitors or inducers
* Diagnosis of any second malignancy within 3 years prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-09-03 (Actual); Primary Completion 2014-11-06 (Actual); Study Completion 2014-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- United States (5):
  - Anschutz Inpatient Pavilion, Aurora, Colorado
  - University of Colorado Cancer Center, Aurora, Colorado
  - University of Colorado Denver, CTO (CTRC), Aurora, Colorado
  - University of Rochester Investigational Drug Pharmacy, Rochester, New York
  - University of Rochester, Rochester, New York

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8641019&StudyName=%EF%82%86%0APhase%201%2F2%20Study%20Of%20Pf-03084014%20In%20Combination%20With%20Gemcitabine%20And%20Nab-paclitaxel%20In%20Patients%20With%20Previously%20Untreated%20Metastatic%20Pancreatic%20Ductal%20Adenocarcinoma%0A

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study planned to include 2 phases: Phase 1 (dose-finding phase) followed by Phase 2 (randomized phase). Due to early termination of the study, only 3 participants were enrolled in Phase 1 and Phase 2 was not conducted.
Groups:
- PF-03084014+Nab-Paclitaxel+Gemcitabine: PF-03084014 was administered twice daily (BID) orally via tablets at a starting dose of 100 milligrams (mg). Nab-paclitaxel (nab-P) and gemcitabine (GEM) were administered intravenously at a starting dose of 125 mg/square meter (m^2) and 1000 mg/m^2, respectively. Decisions to escalate, de-escalate or stay at the same dose were made based on the number of dose-limiting toxicities (DLTs) observed. In any case, PF-03084014 dose was not to exceed 150 mg BID and nab-P and GEM were not to exceed 125 mg/m^2 and 1000 mg/m^2, respectively.
Period: Overall Study
Arm/Group | PF-03084014+Nab-Paclitaxel+Gemcitabine
Started | 3
Completed | 0
Not Completed | 3
Not completed — Symptomatic deterioration | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | PF-03084014+Nab-Paclitaxel+Gemcitabine
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLTs) in Cycle 1
Description: DLT was defined as any of the following events occurring during the first cycle of treatment and considered at least possibly-related to study medication: any Grade 3 or 4 clinically-relevant non-hematologic and/or hematologic toxicity, delay of more than 2 weeks in receiving the next scheduled cycle due to persisting treatment-related toxicities.
Time Frame: Cycle 1 (28 days)
Population: All enrolled participants who received study treatment and who either experienced DLT during the first cycle, or completed the 1-cycle observation period, were considered evaluable for DLT. Only 2 of the 3 participants were evaluable for DLTs.
Measure: Number; unit: participants
Groups:
- PF-03084014 + Nab-Paclitaxel + Gemcitabine: PF-03084014 was administered twice daily (BID) orally via tablets at a starting dose of 100 milligrams (mg). Nab-paclitaxel (nab-P) and gemcitabine (GEM) were administered intravenously at a starting dose of 125 mg/square meter (m^2) and 1000 mg/m^2, respectively. Decisions to escalate, de-escalate or stay at the same dose were made based on the number of dose-limiting toxicities (DLTs) observed. In any case, PF-03084014 dose was not to exceed 150 mg BID and nab-P and GEM were not to exceed 125 mg/m^2 and 1000 mg/m^2, respectively.
Arm/Group | PF-03084014 + Nab-Paclitaxel + Gemcitabine
Number analyzed (Participants) | 2
participants | 2

2. Primary Outcome: Overall Survival (OS) in Phase 2
Description: Overall survival was the duration from randomization to death. For participants who are alive, overall survival was censored at the last contact.
Time Frame: From start of study treatment, collected every 3 months until death (up to 5 years)
Population: All randomized participants in Phase 2 were to be analyzed for OS. However, since Phase 2 was not carried out due to early termination, no subjects were analyzed for OS.
Arm/Group | PF-03084014 + Nab-Paclitaxel + Gemcitabine
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Adverse Events (AEs) by Seriousness and Relationship to Treatment in Phase 1
Description: Counts of participants who had treatment-emergent adverse events (TEAEs), defined as newly occurring or worsening after first dose. Relatedness to study drug was assessed by the investigator (Yes/No). Participants with multiple occurrences of an AE within a category were counted once within the category. Severity was graded by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE). Grade 1=mild, Grade 2=moderate, Grade 3=Severe or medically significant but not immediately life-threatening, Grade 4=life-threatening.
Time Frame: Baseline up to 28-35 days post last administration of study drug
Population: All enrolled participants in Phase 1 who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-03084014 + Nab-Paclitaxel + Gemcitabine
Number analyzed (Participants) | 3
participants
  All-causality TEAEs | 3
  Treatment-related TEAEs | 3
  Grade 3 or 4 TEAEs | 3

4. Secondary Outcome: Number of Participants With Adverse Events (AEs) by Seriousness and Relationship to Treatment in Phase 2
Description: as for outcome 3
Time Frame: Baseline up to 28-35 days post last administration of study drug
Population: No participants were analyzed since Phase 2 was not performed.
Arm/Group | PF-03084014 + Nab-Paclitaxel + Gemcitabine
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Phase 1
Description: Following parameters were analyzed for laboratory examination: hematology (hemoglobin, platelet count, white blood cell count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes); blood chemistry (urea, creatinine, glucose, calcium, sodium, potassium, chloride, magnesium, phosphate, aspartate aminotransferase, alanine aminotransferase, total bilirubin, alkaline phosphatase, uric acid); urinalysis (protein, blood, microscopy[if urine tested positive for blood or protein]).
Time Frame: Screening; Cycle 1 Days 1, 8, 15, 22; up to 28-35 days post last administration of study drug
Population: All participants who received any study treatment.
Measure: Number; unit: participants
Arm/Group | PF-03084014 + Nab-Paclitaxel + Gemcitabine
Number analyzed (Participants) | 3
participants | 3

6. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Phase 2
Description: as for outcome 5
Time Frame: Screening; Days 1, 8, 15 of each cycle; up to 28-35 days post last administration of study drug
Population: Due to early termination, Phase 2 was not performed and thus no participants were included in this analysis.
Arm/Group | PF-03084014 + Nab-Paclitaxel + Gemcitabine
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs at Phases 1 and 2
Description: Following parameters were analyzed for examination of vital signs: systolic and diastolic blood pressure, heart rate, weight and body surface area.
Time Frame: Baseline up to 28-35 days after treatment discontinuation
Population: All enrolled participants in Phase 1, or all randomized participants in Phase 2, who received at least 1 dose of study medication. Due to early termination of the study, vital sign evaluations were not performed.
Arm/Group | PF-03084014 + Nab-Paclitaxel + Gemcitabine
Number analyzed (Participants) | 0

8. Secondary Outcome: Number of Participants With Worsening QTc Results in Phase 1
Description: Triplicate 12-lead electrocardiogram (ECG) measurements (each recording separated by approximately 2 minutes) were performed and average was calculated. The time corresponding to beginning of depolarization to repolarization of the ventricles (QT interval) were corrected for heart rate (QTc) using Fridericia (QTcF) and Bazett (QTcB) formulas. Any change from baseline in QTc was considered as worsening in ECG and was classified accordingly to the Common Terminology Criteria (CTC) grade. Grading was as follows: prolonged QTc of 450 to 480 milliseconds (msec)=Grade 1, 481 to 500 msec=Grade 2, more than or equal to (>=) 501 msec on at least 2 seperate ECGs=Grade 3, >=501 or more than (>) 60 msec change from baseline and Torsade de pointes or polymorphic ventricular tachycardia or signs of serious arrhythmia=Grade 4.
Time Frame: Screening, Cycle 1 Days 3 and 22, Cycles 2 and 3 Day 1, end of treatment
Population: All enrolled participants in Phase 1 who had at least 1 ECG assessment after receiving PF-03084014.
Measure: Number; unit: participants
Arm/Group | PF-03084014 + Nab-Paclitaxel + Gemcitabine
Number analyzed (Participants) | 3
participants | NA — Results were all outside of the toxicity range and could not be evaluated.

9. Secondary Outcome: Number of Participants With Worsening QTc Results in Phase 2
Description: as for outcome 8
Time Frame: Screening, Cycle 1 Days 1 and 22, Cycles 2 and 3 Day 1, end of treatment
Population: Due to early termination, Phase 2 was not performed and thus no participants were analyzed for this outcome measure.
Arm/Group | PF-03084014 + Nab-Paclitaxel + Gemcitabine
Number analyzed (Participants) | 0

10. Secondary Outcome: Area Under the Concentration-time Curve (AUC) for PF-03084014, Nab-P and Gemcitabine in Phase 1
Description: AUC included AUC from time 0 extrapolated to infinite time (AUCinf), AUC from time 0 to end of dosing interval (AUCtau, tau=12 hours), and AUC from time 0 to last measured concentration (AUClast).
Time Frame: PF-03084014: Cycle 1 Days 3, 15, 22; Day 1 of subsequent cycles; and end of treatment. nab-P: Cycle 1 Days 1-3 and 15-17. Gemcitabine: Cycle 1 Days 1 and 15.
Population: All treated participants who had at least 1 of the pharmacokinetic (PK) parameters of interest of any of the study drugs. n=number of evaluable participants for that parameter at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | PF-03084014 + Nab-Paclitaxel + Gemcitabine
Number analyzed (Participants) | 3
nanogram*hour/milliliter (ng*hr/mL)
  AUClast for PF-03084014 on Day 3 (n=3) | 1122 (913)
  AUClast for PF-03084014 on Day 15 (n=1) | 1770 (NA) — The Geometric Coefficient of Variation is not calculable as there was one evaluable participant.
  AUCinf for nab-paclitaxel on Day 1 (n=3) | 5774 (11)
  AUClast for nab-paclitaxel on Day 1 (n=3) | 5185 (9)
  AUCinf for nab-paclitaxel on Day 15 (n=1) | 5050 (NA) — The Geometric Coefficient of Variation is not calculable as there was one evaluable participant.
  AUClast for nab-paclitaxel on Day 15 (n=1) | 4600 (NA) — The Geometric Coefficient of Variation is not calculable as there was one evaluable participant.
  AUCinf for gemcitabine on Day 1 (n=3) | 5316 (172)
  AUClast for gemcitabine on Day 1 (n=3) | 5262 (176)
  AUCinf for gemcitabine on Day 15 (n=1) | 2510 (NA) — The Geometric Coefficient of Variation is not calculable as there was one evaluable participant.
  AUClast for gemcitabine on Day 15 (n=1) | 2500 (NA) — The Geometric Coefficient of Variation is not calculable as there was one evaluable participant.

11. Secondary Outcome: Area Under the Concentration-time Curve (AUC) for PF-03084014, Nab-P and Gemcitabine in Phase 2
Description: AUC included AUC from time 0 extrapolated to infinite time (AUCinf), AUC from time 0 to end of dosing interval (AUCtau), and AUC from time 0 to last measured concentration (AUClast).
Time Frame: Cycle 1 Day 1 till end of last cycle
Population: As Phase 2 was not performed, no participants were analyzed for this outcome measure.
Arm/Group | PF-03084014 + Nab-Paclitaxel + Gemcitabine
Number analyzed (Participants) | 0

12. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for PF-03084014, Nab-P and GEM in Phase 1
Time Frame: as for outcome 10
Population: All treated participants who had at least 1 of the PK parameters of interest of any of the study drugs. n=number of evaluable participants for that parameter at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | PF-03084014 + Nab-Paclitaxel + Gemcitabine
Number analyzed (Participants) | 3
nanogram/milliliter (ng/mL)
  Cmax for PF-03084014 on Day 3 (n=3) | 527.3 (710)
  Cmax for PF-03084014 on Day 15 (n=1) | 943.0 (NA) — The Geometric Coefficient of Variation is not calculable as there was one evaluable participant.
  Cmax for nab-paclitaxel on Day 1 (n=3) | 6023 (6)
  Cmax for nab-paclitaxel on Day 15 (n=1) | 5140 (NA) — The Geometric Coefficient of Variation is not calculable as there was one evaluable participant.
  Cmax for gemcitabine on Day 1 (n=3) | 10760 (212)
  Cmax for gemcitabine on Day 15 (n=1) | 3620 (NA) — The Geometric Coefficient of Variation is not calculable as there was one evaluable participant.

13. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for PF-03084014, Nab-P and GEM in Phase 2
Time Frame: Cycle 1 Day 1 till end of last cycle
Population: As Phase 2 was not performed, no participants were analyzed for this outcome measure.
Arm/Group | PF-03084014 + Nab-Paclitaxel + Gemcitabine
Number analyzed (Participants) | 0

14. Secondary Outcome: Systemic Clearance (CL) of Nab-paclitaxel in Phase 1
Time Frame: Cycle 1 Days 1-3, and 15-17
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter (L)/hour (hr)
Arm/Group | PF-03084014 + Nab-Paclitaxel + Gemcitabine
Number analyzed (Participants) | 3
liter (L)/hour (hr)
  Day 1 (n=3) | 37.88 (25)
  Day 15 (n=1) | 38.60 (NA) — The Geometric Coefficient of Variation is not calculable as there was one evaluable participant.

15. Secondary Outcome: Systemic Clearance (CL) of Gemcitabine in Phase 1
Time Frame: Cycle 1 Days 1 and 15
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter (L)/minute (min)
Arm/Group | PF-03084014 + Nab-Paclitaxel + Gemcitabine
Number analyzed (Participants) | 3
liter (L)/minute (min)
  Day 1 (n=3) | 5.434 (165)
  Day 15 (n=1) | 8.160 (NA) — The Geometric Coefficient of Variation is not calculable as there was one evaluable participant.

16. Secondary Outcome: Systemic Clearance (CL) of PF-03084014, Nab-P and GEM in Phase 2
Time Frame: Cycle 1 Day 1 till end of last cycle
Population: As Phase 2 was not performed, no participants were analyzed for this outcome measure.
Arm/Group | PF-03084014 + Nab-Paclitaxel + Gemcitabine
Number analyzed (Participants) | 0

17. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) for PF-03084014, Nab-P and GEM in Phase 1
Time Frame: as for outcome 10
Population: as for outcome 12
Measure: Median (Full Range); unit: hours
Arm/Group | PF-03084014 + Nab-Paclitaxel + Gemcitabine
Number analyzed (Participants) | 3
hours
  Tmax of PF-03084014 on Day 3 (n=3) | 1.23 [0.517 to 4.13]
  Tmax of PF-03084014 on Day 15 (n=1) | 0.900 [NA to NA] — Range is not applicable as there is only a single evaluable participant at this time point.
  Tmax of nab-paclitaxel on Day 1 (n=3) | 0.550 [0.517 to 0.583]
  Tmax of nab-paclitaxel on Day 15 (n=1) | 0.217 [NA to NA] — Range is not applicable as there is only a single evaluable participant at this time point.
  Tmax of gemcitabine on Day 1 (n=3) | 0.517 [0.250 to 0.533]
  Tmax of gemcitabine on Day 15 (n=1) | 0.350 [NA to NA] — Range is not applicable as there is only a single evaluable participant at this time point.

18. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) for PF-03084014, Nab-P and GEM in Phase 2
Time Frame: Cycle 1 Day 1 till end of last cycle
Population: As Phase 2 was not performed, no participants were analyzed for this outcome measure.
Arm/Group | PF-03084014 + Nab-Paclitaxel + Gemcitabine
Number analyzed (Participants) | 0

19. Secondary Outcome: Volume of Distribution at Steady State (Vss) for Nab-P and GEM in Phase 1
Time Frame: Cycle 1 (Days 1 and 15 for gemcitabine; Days 1-3 and 15-17 for nab-paclitaxel)
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | PF-03084014 + Nab-Paclitaxel + Gemcitabine
Number analyzed (Participants) | 3
liters
  Vss of nab-paclitaxel on Day 1 (n=3) | 64.46 (6)
  Vss of nab-paclitaxel on Day 15 (n=1) | 60.80 (NA) — The Geometric Coefficient of Variation is not calculable as there was one evaluable participant.
  Vss of gemcitabine on Day 1 (n=3) | 61.76 (186)
  Vss of gemcitabine on Day 15 (n=1) | 201.0 (NA) — The Geometric Coefficient of Variation is not calculable as there was one evaluable participant.

20. Secondary Outcome: Volume of Distribution at Steady State (Vss) for PF-03084014, Nab-P and GEM in Phase 2
Time Frame: Cycle 1 Day 1 till end of last cycle
Population: As Phase 2 was not performed, no participants were analyzed for this outcome measure.
Arm/Group | PF-03084014 + Nab-Paclitaxel + Gemcitabine
Number analyzed (Participants) | 0

21. Secondary Outcome: Plasma Decay Half-life (t1/2) for Nab-P and GEM in Phase 1
Time Frame: Cycle 1 (Days 1 and 15 for gemcitabine; Days 1-3 and 15-17 for nab-paclitaxel)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PF-03084014 + Nab-Paclitaxel + Gemcitabine
Number analyzed (Participants) | 3
hours
  t1/2 of nab-paclitaxel on Day 1 (n=3) | 2.500 (0.26851)
  t1/2 of nab-paclitaxel on Day 15 (n=1) | 2.030 (NA) — The Standard Deviation is not calculable as there was one evaluable participant.
  t1/2 of gemcitabine on Day 1 (n=3) | 0.2813 (0.14838)
  t1/2 of gemcitabine on Day 15 (n=1) | 0.2230 (NA) — The Standard Deviation is not calculable as there was one evaluable participant.

22. Secondary Outcome: Plasma Decay Half-life (t1/2) for PF-03084014, Nab-P and GEM in Phase 2
Time Frame: Cycle 1 Day 1 till end of last cycle
Population: As Phase 2 was not performed, no participants were analyzed for this outcome measure.
Arm/Group | PF-03084014 + Nab-Paclitaxel + Gemcitabine
Number analyzed (Participants) | 0

23. Secondary Outcome: Number of Participants With Objective Response (OR) in Phase 1
Description: Number of participants with objective response based on assessment of complete response (CR) or partial response (PR) according to Response Evaluation Criteria In Solid Tumors (RECIST).
  CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis less than (<) 10 mm). No new lesions. PR was defined as more than or equal to (>=) 30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions.
Time Frame: Screening till 28-35 days post last administration of study drug
Population: All enrolled participants in Phase 1 who were eligible for enrollment, received study treatment, had measurable disease and adequate baseline assessments, and had at least 1 on-study tumor assessment, were considered evaluable for response. Only 1 participant was evaluable for OR in Phase 1.
Measure: Number; unit: participants
Arm/Group | PF-03084014 + Nab-Paclitaxel + Gemcitabine
Number analyzed (Participants) | 1
participants | 0

24. Secondary Outcome: Number of Participants With Objective Response (OR) in Phase 2
Description: as for outcome 23
Time Frame: Screening till 28-35 days post last administration of study drug
Population: No participants were analyzed for this outcome measure as Phase 2 was not done.
Arm/Group | PF-03084014 + Nab-Paclitaxel + Gemcitabine
Number analyzed (Participants) | 0

25. Secondary Outcome: Duration of Response (DR) for Phases 1 and 2
Description: Duration of response (DR) defined as the difference in days between the first date criteria for progression occurred or the participant died due to any cause and the first date that criteria for a PR or CR were met. DR calculated as (months) = (progression/death date - first date of OR + 1) divided by 30.4. CR: disappearance of all target lesions. PR: at least 30% decrease in the sum of diameters of target lesions.
Time Frame: Baseline, every 8 weeks until disease progression or unacceptable toxicity (up to 5 years)
Population: No participants were analyzed for this outcome measure as there were no participants with OR in Phase 1 and Phase 2 was not done.
Arm/Group | PF-03084014 + Nab-Paclitaxel + Gemcitabine
Number analyzed (Participants) | 0

26. Secondary Outcome: 1-year and 2-year OS in Phase 2
Description: as for outcome 2
Time Frame: From start of study treatment, collected every 3 months until death (up to 5 years)
Population: as for outcome 2
Arm/Group | PF-03084014 + Nab-Paclitaxel + Gemcitabine
Number analyzed (Participants) | 0

27. Secondary Outcome: Progression-free Survival (PFS) in Phase 2
Description: PFS was defined as the time from the date of first dose to the date of the first documentation of objective tumor progression or death on study due to any cause, whichever occurred first. PFS (in months) was calculated as (first event date - date of randomization +1) divided by 30.4.
Time Frame: From start of study treatment, collected every 3 months until death (up to 5 years)
Population: All randomized participants in Phase 2 were to be analyzed for PFS. However, since Phase 2 was not carried out due to early termination, no subjects were analyzed for PFS.
Arm/Group | PF-03084014 + Nab-Paclitaxel + Gemcitabine
Number analyzed (Participants) | 0

28. Secondary Outcome: Brief Pain Inventory-Short Form (BPI-sf) Score - Phase 2
Description: BPI-sf is an 11-item self-report questionnaire that is designed to assess the severity and impact of pain on daily functions. BPI-sf are 4 questions that assess pain intensity (worst, least, average, right now) and 7 questions that assess impact of pain on daily functions (general activity, mood, walking ability, normal work, relations with other people, sleep, enjoyment of life). Each question is answered on a scale ranging from 0 to 10; '0=No pain and 10=Pain as bad as you can imagine'. Measure can be scored by item, with lower scores being indicative of less pain or pain interference.
Time Frame: Day 1 of Cycle 1 and subsequent cycles; end of treatment
Population: As Phase 2 was not performed due to early termination, there were no participants to analyse for this outcome measure.
Arm/Group | PF-03084014 + Nab-Paclitaxel + Gemcitabine
Number analyzed (Participants) | 0

29. Secondary Outcome: Change From Baseline in European Quality of Life Questionnaire (EQ-5D) - Phase 2
Description: EQ-5D: 6-item participant rated questionnaire to assess health-related quality of life in terms of a single utility score. There were 2 components: a Health State Profile and a Visual Analog Scale. Published weights are available that allow for the creation of a single summary score. Overall scores range from 0-1, with low scores representing a higher level of dysfunction.
Time Frame: Baseline till end of treatment
Population: As Phase 2 was not performed due to early termination, there were no participants to analyse for this outcome measure.
Arm/Group | PF-03084014 + Nab-Paclitaxel + Gemcitabine
Number analyzed (Participants) | 0

30. Secondary Outcome: European Organization for Research and Treatment of Cancer, Quality of Life Questionnaire (EORTC QLQ-C30) - Phase 2
Description: EORTC QLQ-C30: included functional scales (physical, role, cognitive, emotional, and social), global health status, symptom scales (fatigue, pain, nausea/vomiting) and single items (dyspnoea, appetite loss, insomnia, constipation/diarrhea and financial difficulties). Most questions used 4-point scale (1 'Not at all' to 4 'Very much'; 2 questions used 7-point scale (1 'very poor' to 7 'Excellent'). Scores averaged, transformed to 0-100 scale; higher score=better level of functioning or greater degree of symptoms.
Time Frame: Baseline till end of treatment
Population: As Phase 2 was not performed due to early termination, there were no participants to analyse for this outcome measure.
Arm/Group | PF-03084014 + Nab-Paclitaxel + Gemcitabine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline through and including 28 calendar days after the last administration of the investigational product.
Arm/Group | PF-03084014+Nab-Paclitaxel+Gemcitabine
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-03084014+Nab-Paclitaxel+Gemcitabine (N=3)
Vomiting (Gastrointestinal disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-03084014+Nab-Paclitaxel+Gemcitabine (N=3)
Ascites (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Chills (General disorders) | 1
Fatigue (General disorders) | 3
Mucosal inflammation (General disorders) | 1
Candida infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
Due to early termination of the study, only 3 participants were enrolled. Phase 2 was not carried out. As such, there is limited data for Phase 1 and no data for Phase 2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.